CLINICAL TRIAL: NCT04100382
Title: Implant Stability in Laser Treated Surface vs SLA Treated Short Implants (Randomized Clinical Trial)
Brief Title: Laser Treated vs SLA Treated Short Implants in Terms of Stability.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Alaa Diab, Principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1719
Record Dates: First submitted 2019-09-13; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Will Laser Treated Dental Implants Improve Stability Early Healing
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser and SLA implants (Experimental): Surgical placement of short implants in maxillary posterior teeth with Laser surface treated and SLA surface treated dental implants
  Interventions: Device: Laser and SLA

INTERVENTIONS:
Device: Laser and SLA — Patients will be randomized into two groups, control group for SLA implants, and study group will receive the Laser treated implants. Implants will be placed classically in the posterior maxillary region and their stability will be measured by ISQ device at the placement. Measurements will be taken again at 2, 4, 6, 8 , 10 and 12 weeks.

SUMMARY:
Laser treated short dental implants will be placed in a posterior atrophic ridge with only 8-10 mm available bone height. Their stability will be measured through a period of 12 weeks. They will be compared to the stability of SLA treated Short dental implants placed in the same situations.

DETAILED DESCRIPTION:
Laser treated short dental implants will be placed in a posterior atrophic ridge with only 8-10 mm available bone height. Their stability will be measured through a period of 12 weeks. They will be compared to the stability of SLA treated Short dental implants placed in the same situations.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients with Edentulous posterior maxillae with insufficient ridge for placement of standard length dental implant, but allowing placement of short 8mm dental implant.

  * Males and females.

Exclusion Criteria:

* • Heavy smokers more than 20 cigarettes per day.

  * Patients with systemic disease that may affect normal healing.
  * Psychiatric problems
  * Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site
  * Patients suffering from immunodeficiency, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.
  * Intraoral soft and hard tissue pathology.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Rate of change in implant stability at base line, 2,4,8, 12 weeks | 3 months
  measuring implant stability with resonance frequency analysis device using implant stability quotation (ISQ) that measures the stiffness and deflection of implant bone complex.